CLINICAL TRIAL: NCT03958604
Title: Prospective Post Market Pilot Study to Evaluate the Effectiveness of Burst Spinal Cord Stimulation in the Treatment of Discogenic Low Back Pain
Brief Title: Burst Neurostimulation for Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL 67172.091.18
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2021-12

CONDITIONS: Discogenic Pain; Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Burst neurostimulation for discogenic low back pain. If this fails to provide pain relief of at least 50%, tonic stimulation targeting the DRG will be the second treatment potential. Follow-up during one year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Burst Spinal Cord Neurostimulation (Experimental): Burst spinal cord stimulation. When this fails, tonic stimulation targeting the DRG wil be applied
  Interventions: Procedure: Neurostimulation

INTERVENTIONS:
Procedure: Neurostimulation — Spinal cord stimulation with burst modality for discogenic low back pain
  Other Names: spinal cord burst stimulation; spinal cord stimulation; ProdigyTM Abbott Laboratories; ProclaimTM Abbott Laboratories

SUMMARY:
The purpose of this prospective post market pilot study is to evaluate the effect of Burst Spinal Cord Stimulation(B-SCS) in the management of chronic discogenic pain in subjects who are refractory to other available treatments. Selected subjects will not be suitable candidates for lumbar spinal surgery and will meet the standard selection process for SCS as routinely utilized in the study centers. Results from this pilot study will inform current clinical practice and future comparative studies in this specific population. Eligible subjects for B-SCS will be asked to participate in this study. If they decide to participate, they will be treated with the Prodigy TM and Proclaim TM (Abbott Laboratories) SCS system and prospectively followed for 12 months following implantation.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center, post-market, pilot study to collect data on back pain relief, subject satisfaction, quality of life, physical functioning and safety. Chronic discogenic pain(CDP) suffering patients will be followed for 12 months with follow-up visits at 3, 6, and 12 months. In line with standard practice the system will be implanted in two stages. The first stage is the Trial Burst spinal cord Neurostimulation (TBNS) phase during which epidural leads are implanted and temporarily tunnelled to an external trial stimulation device. Subjects will then utilize the temporary system for a period in line with usual practice (typically 10-14 days). If, at the end of this TBNS phase a reduction of ≥50% is achieved the device will be permanently implanted (the second stage) and subjects will be followed-up during 12 months. Patients who do not have at least 50% pain relief during TBNS will receive a Trial Tonic Neurostimulator(TTNS) targeting the dorsal root ganglion(DRG). Similarly, these patients will be followed-up during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to comply with the follow-up schedule and protocol
* Subject is able to provide written informed consent
* Chronic low back pain of at least 6 months
* History consistent with discogenic low back pain (e.g. Pain produced on lumbar motion, significant functional limitation in sitting duration and tolerance)
* Subject has a negative test block of facet joints in the sacroiliac joint.
* Neurologic exam without marked motor deficit.
* Definite/Highly Probable/Discogenic Pain as confirmed by provocative discography according to International Association for the Study of Pain (IASP/ISIS) guidelines
* Low Back Pain intensity should be 6 or higher measured on a Numeric Pain Rating Scale(NPRS) at baseline
* Meets all the inclusion criteria for the implantation of a neurostimulation system as typically utilized in the study center
* Subject has been screened by a multi-disciplinary panel including a psychologist and deemed suitable for implantation

Exclusion Criteria:

* Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study
* Escalating or changing pain condition within the past month as evidenced by investigator examination
* Body Mass Index ≥35
* Subject has had injection therapy or radiofrequency treatment for their low back pain within the past 3 months
* Subject currently has an active implantable device including Internal Cardioverter Defibrillator(ICD), pacemaker, spinal cord stimulator, or intrathecal drug pump
* Subject is unable to operate the device
* Severe disc degeneration at the affected level as evidenced by >50% disc height loss on plain anteroposterior and lateral lumbar radiographs of ComputoTomography (CT)/Magnetic Resonance Imaging(MRI).
* Extruded or sequestered herniated nucleus pulposus at the affected level(s).
* Previous lumbar back surgery (e.g. Laminectomy, discectomy or fusion) at the affected level(s)
* Moderate to severe spinal stenosis due to osteophyte and/or ligamentous overgrowth as evidenced by MRI or CT in the previous 6 months
* Moderate to severe endplate degenerative changes at the affected levels Grade 1-2 spondylolisthesis
* Previous Neurostimulation(SCS) therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain severity | 1 year
  Pain severity, assessed by an 11 point (0-10) numerical pain rating scale 0=no pain, 10 very severe pain

SECONDARY OUTCOMES:
Treatment satisfaction | 1 year
  Patient's Global Impression of Change, a 7-point Likert scale ( 1 =very much improved and 7 is very much worse
Disability | 1 year
  Physical function will be assessed using the Oswestry Disability Index
Quality of Life utility score | 1 year
  EuroQol-5D-5L
Safety; Serious and Adverse events | 1 year
  Safety will be monitored by the collection and reporting of device related adverse events, device related serious adverse events and any unanticipated serious adverse events (regardless of device relatedness).
Pain type | 1 year
  PainDETECT® questionnaire which is designed to differentiate between neuropathic and non-neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Kallewaard, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate hospital Pain Management Centre Velp, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courtney P, Espinet A, Mitchell B, Russo M, Muir A, Verrills P, Davis K. Improved Pain Relief With Burst Spinal Cord Stimulation for Two Weeks in Patients Using Tonic Stimulation: Results From a Small Clinical Study. Neuromodulation. 2015 Jul;18(5):361-6. doi: 10.1111/ner.12294. Epub 2015 Apr 16. PMID 25879884
- [Background] Kallewaard JW, Terheggen MA, Groen GJ, Sluijter ME, Derby R, Kapural L, Mekhail N, van Kleef M. 15. Discogenic low back pain. Pain Pract. 2010 Nov-Dec;10(6):560-79. doi: 10.1111/j.1533-2500.2010.00408.x. Epub 2010 Sep 6. PMID 20825564
- [Derived] Mons MR, Chapman KB, Terwiel C, Joosten EA, Kallewaard JW. Burst Spinal Cord Stimulation as Compared With L2 Dorsal Root Ganglion Stimulation in Pain Relief for Nonoperated Discogenic Low Back Pain: Analysis of Two Prospective Studies. Neuromodulation. 2024 Jan;27(1):172-177. doi: 10.1016/j.neurom.2023.04.464. Epub 2023 May 16. PMID 37191612
- [Derived] Mons MR, Chapman KB, Terwiel C, Joosten EA, Kallewaard JW. A prospective study of BurstDR spinal cord stimulation for non-operated discogenic low back pain. Pain Pract. 2023 Mar;23(3):234-241. doi: 10.1111/papr.13181. Epub 2022 Nov 23. PMID 36373868